CLINICAL TRIAL: NCT00116571
Title: A Phase II Randomized, Sham-Controlled, Double-Blind, Dose-Finding Study to Assess the Efficacy and Safety of Transurethral Photodynamic Therapy With Lemuteporfin in Subjects With Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia
Brief Title: Photodynamic Therapy (PDT) for Lower Urinary Tract Symptoms (PLUS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: QLT Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BPH 003
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Last update posted 2006-10-03 (Estimated); Status verified 2006-05

CONDITIONS: Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia (BPH); Photodynamic Therapy (PDT); Lower Urinary Tract Symptoms (LUTS)
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — lemuteporfin; Injections

INTERVENTIONS:
Drug: Lemuteporfin for injection
Device: Transurethral drug delivery system
Device: Transurethral light delivery system

SUMMARY:
The purpose of this study is to determine if transurethral photodynamic therapy with lemuteporfin has a therapeutic effect on lower urinary tract symptoms due to an enlarged prostate.

Photodynamic therapy (known as "PDT") is a treatment that uses light to make a drug work. This means the drug is "light-activated". Light-activated drugs do not work until a certain color of light shines on the drug. When the drug and the light combine, they react together to destroy tissue.

This study is investigating PDT with lemuteporfin as a possible treatment for an enlarged prostate. PDT with lemuteporfin may destroy overgrown prostate tissue and help urinary symptoms go back to normal.

DETAILED DESCRIPTION:
This is a multi-center, randomized, sham-controlled, double-blind, dose-finding study in parallel groups of subjects with lower urinary tract symptoms (LUTS) due to benign prostatic hyperplasia (BPH). All subjects will receive a fixed dose of lemuteporfin injected transurethrally into the prostate followed by transurethral application of either one of three active light doses or a sham light dose. Subjects will be followed for safety and efficacy for a minimum of three months to a maximum of 12 months. The primary study endpoint will be the change from baseline in AUA SI score at three months.

ELIGIBILITY:
Inclusion Criteria:

* Men 21 years of age and older.
* Subjects with LUTS due to BPH with AUA SI scores of 13 and over and Qmax between 5 and 15 mL/sec.
* Subjects with urethral treatment length of at least 25 mm.

Exclusion Criteria:

* Subjects who have had previous minimally invasive or surgical treatment for BPH.
* Subjects who have unsuitable prostate dimensions.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2005-05; Study Completion 2006-12

PRIMARY OUTCOMES:
The change from baseline in American Urological Association Symptom Index (AUA SI) score at the Month 3 visit

SECONDARY OUTCOMES:
Responder rate
Change from baseline in Qmax
Change from baseline in post-void residual (PVR)
Shifts from baseline in subject responses to the BPH Quality of Life Impact Assessment
Safety outcomes: adverse events, clinical laboratory tests, vital signs, dysuria, and Male Sexual Health Questionnaire (MSHQ)

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Boniface, PhD, Study Director — QLT Inc.
Locations (9):
- United States (8):
  - San Bernardino Urological Associates, San Bernardino, California
  - Regional Urology, LLC, Shreveport, Louisiana
  - Drs Werner, Murdock & Francis PA Urology Associates, Greenbelt, Maryland
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - AccuMed Research Associates, Garden City, New York
  - Duke University Medical Center, Durham, North Carolina
  - Urology San Antonio Research, PA, San Antonio, Texas
  - Devine Tidewater Urology, Virginia Beach, Virginia
- Can-Med Clinical Research Inc, Victoria, British Columbia, Canada